CLINICAL TRIAL: NCT02952625
Title: An Exploratory Study to Assess the Feasibility of Incorporating PET/MR in the Radiotherapy Pathway of Patients With Head and Neck Cancer and Guide Adaptive Dose Escalation
Brief Title: PET/MR in Radiotherapy for Head and Neck Cancer Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RJ116/N013
Record Dates: First submitted 2016-10-25; First posted 2016-11-02 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Head and Neck Cancer
Keywords: PET/MRI
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm imaging study (Other): Single arm study: all patients have 2 PET/MR scans in the radiotherapy treatment position
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — Single arm Imaging (PET/MR) study

SUMMARY:
This is a pilot non-intervention study that aims to introduce PET/MRI, a state of the art new imaging technique, into the radiotherapy treatment pathway of patients with head and neck cancer. Ultimately the investigators aim to establish appropriate scanning and image registration protocols, to allow progression to a randomized trial of adaptive radiotherapy dose escalation. The latter is thought to potentially improve outcomes in this group.

Ten patients with squamous cell carcinoma (SCC) of the oropharynx, hypopharynx and larynx, planned for radical treatment with radiotherapy (+/-chemotherapy), will be recruited. Study participants will have two PET/MRI scans, with the radiotherapy immobilization devices in situ. The first will be done prior to the start of radiotherapy, the second half way through treatment.

Image quality will be assessed by comparing to standard diagnostic scans and different registration methods will be compared to establish the best way of incorporating PET/MR image data into the radiotherapy planning system. Patient tolerability and workflow considerations will also be qualitatively assessed. Furthermore, a planning study will be conducted to establish relevant treatment protocols for a subsequent dose escalation trial.

PET/MRI is an exciting new technology with a lot of potential in the context of adaptive radiotherapy dose escalation. Within this pilot study the investigators aim to address the technical challenges of using it in this context prior to proceeding to a randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Written, voluntary, informed consent
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Life expectancy > 12 months
* Histologically proven SCC of the oropharynx, hypopharynx and larynx
* Radical radiotherapy +/- chemotherapy indicated as the primary treatment modality
* Visible disease (>1cm) at the primary site on any imaging modality performed within 4 weeks of starting radiotherapy treatment
* Staging PET/CT and diagnostic MRI of the head and neck images need to be available for comparison.
* Adequate organ function and absence of other major concurrent illness, allowing the patient to tolerate scanning regime

Exclusion Criteria:

* Inability to provide informed consent
* Impaired renal function (serum creatinine of > 200)
* Severely impaired liver function
* Patients with allergies or contra-indications to the radio-tracer and/or contrast agent used in the study
* Severe claustrophobia or inability to tolerate PET or MRI scans
* General contra-indications to MRI, as defined in MRI safety departmental protocols
* Serious inter-current conditions or other non-malignant illnesses that are uncontrolled or whose control may be affected by participation in this study
* Any patient who has urinary or faecal incontinence
* ECOG Performance Status ≥ 3
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Number of scans where image quality is sufficient to characterise the primary tumour, assessed qualitatively by an experienced radiologist and oncologist | 6 months following study completion
Proportion of patients that tolerated the full scanning protocol, assessed by tailored patient questionnaire | 6 months following study completion

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Guerrero Urbano, Principal Investigator — Guy's & St Thomas' NHS Foundation Trust, London, UK
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No